版本号: \_\_V1.0\_\_

# 版本日期: 2023 年 1 月 30 日

# 知情同意书

**研究名称:** 定坤丹联合复方口服避孕药治疗 PCOS 的有效性及安全性: 一项开放标签、非随机对照临床研究

项目负责人: 李荔 电话: 13631446859

申办者:广东省妇幼保健院

在您决定是否参加这项研究之前,请尽可能仔细阅读以下内容。它可以帮助您了解该项研究以及为何要进行这项研究,研究的程序和期限,参加研究后可能给您带来的益处、风险和不适。如果您愿意,您也可以和您的亲属、朋友一起讨论,或者请医生给予解释,帮助您做出决定。

# 1. 研究背景

多囊卵巢综合征(polycystic ovary syndrome, PCOS)是育龄期女性最常见的妇科内分泌紊乱疾病,患病率约为 5%~10%。PCOS 不但会影响妇女的生殖功能,且增加妇女的代谢障碍(例如:腹型肥胖、血脂异常、血糖稳态受损)和罹患心血管疾病的风险。其次,PCOS 妇女的妊娠相关并发症(例如妊娠糖尿病、高血压疾病、早产等)风险明显增加。

PCOS 强调的是个性化的治疗原则,对于无生育要求的女性,主要目标是降低雄激素、调整月经周期、及防治并发症。对于有生育要求的女性,则在此基础上增加诱发排卵、促进生育的治疗。

复方口服避孕药在临床上常用于治疗多囊卵巢综合征,其在帮助建立规律的月经周期和降低雄激素方面有确切的疗效,但停药后病情容易反复发作,且长期服用此药物对患者的肝肾功能及心血管功能不利。

定坤丹由当归、香附、柴胡、川芎等 30 味中药材组成,具有滋补气血、调节月经、提高卵巢功能、疏肝止痛的作用,常用于治疗气血两虚、气滞血瘀所致的妇科疾病,如痛经、月经不调、不孕症、更年期综合征和产后诸虚。目前国内已有一些研究表明,定坤丹联合促排卵药物对 PCOS 不孕的临床效果优于单一使用促排卵药物,使血清 FSH、E2、LH 及 T 等性激素水平降低,并且研究组患者的成熟卵泡直径和子宫内膜厚度都优于对照组,且研究组的妊娠率高于对照组。但国内关于定坤丹治疗 PCOS 的研究仍然很少,且尚无 PCOS 患者使用复方口服避孕药联合定坤丹与单独使用发放口服避孕药的随机对照临床研究。

#### 2. 研究目的

本研究的意义旨在评估复方口服避孕药联合定坤丹在 PCOS 中应用的有效性及安全性,并对比单一使用发放口服避孕药的治疗效果,以期为临床医师根据 PCOS 患者的临床特征,选择更优治疗方案。

## 3. 研究过程

对同意参加本研究的患者,将患者分为研究组(COC+定坤丹)和对照组(COC)。

研究组予以口服优思悦(屈螺酮炔雌醇片(II))治疗,于月经期第1天起按照包装指示服用优思悦(拜耳医药保健有限公司;国药准字:H20140972;规格:屈螺酮 3mg 和炔雌醇(β-环糊精包合物)0.02mg),每日约在同一时间段内服用,连续服用 28 天,停药后月经来潮,在月经第一天开始下一个用药周期。在服用复方口服避孕药的同时加定坤丹浓缩水蜜丸(山西国誉远有限公司,国药准字: Z20059003,规格: 7g/瓶),每次 3.5g,每日两次。

对照组予以口服优思悦(屈螺酮炔雌醇片(II))治疗,于月经期第1天起按照包装指示服用优思悦(拜耳医药保健有限公司;国药准字: H20140972;规格:屈螺酮 3mg 和炔雌醇(β-环糊精包合物)0.02mg),每日约在同一时间段内服用,连续服用 28 天,停药后月经来潮,在月经第一天开始下一个用药周期。两组均连续服药 3 个月为一个疗程。

#### 4. 可能的风险

参与受试者可能出现胃肠道不适,如恶心、呕吐、食欲下降等;或(和)子宫不规则出血;或(和)乳房胀痛。

#### 哪些人不宜参加研究?

- (1) 近3个月内曾服用激素或中药者:
- (2) 有先天性肾上腺皮质增生、库欣综合征、分泌雄激素的肿瘤者;
- (3) 肝肾功能异者;
- (4) 既往有血栓性疾病,动脉或静脉血栓栓塞史者;
- (5) 有重大器质性疾病者。

如果在研究期间您出现任何不适,或病情发生新的变化,或任何意外情况,不管是否与研究有关,均应及时通知您的医生,他/她将对此作出判断并给与适当的医疗处理。

您在研究期间需要按时到医院随访,做一些检查,这些占用您的一些时间, 也可能给您造成麻烦或带来不方便。

#### 5. 受试者收益

通过口服复方口服避孕药+联合坤丹或单独使用复方口服避孕药两组药物,有助于 PCOS 患者的月经周期调节、雄激素的降低、卵巢功能及身体代谢障碍的改善。

#### 6. 相关费用

在诊断和治疗过程中,相关检查费用,如性激素六项、游离睾酮、雄烯二酮、性激素结合球蛋、AMH,空腹血糖、空腹胰岛素、HOMA-IR、同型半胱氨酸、妇科彩超等检查均需个人承担,相关服用药物均需个人承担,可由医保结算。

如出现不良反应时,医生将尽全力预防和治疗由于本研究可能带来的伤害。如果在临床试验中出现不良事件,医学专家委员会将会鉴定其是否与针刺或基础治疗药物有关。申办者将按照我国《药物临床试验质量管理规范》的规定对与试验相关的损害提供治疗的费用及相应的经济补偿)。

对于您同时合并的其他疾病所需的治疗和检查,将不在免费的范围之内。

### 7. 研究记录的保密

如果您决定参加本项研究,您参加试验及在试验中的个人资料均属保密。负责研究医师及其他研究人员将使用您的医疗信息进行研究。这项研究结果发表时,将不会披露您个人的任何资料。

#### 8. 受试者的权利

是否参加试验完全取决于您的自愿。您可以拒绝参加此项试验,或在试验过程中的任何时间退出,这都不会影响对您的治疗或其他方面利益的损失。您可随时了解与本研究有关的信息资料和研究进展,如果您有与本研究有关的问题,或您在研究过程中发生了任何不适与损伤,或有关于本项研究参加者权益方面的问题您可以与研究者或有关人员联系。

#### 个人信息是保密的吗?

您的医疗记录(研究病历/CRF、化验单等)将完整地保存在您所就诊的医院。医生会将化验检查结果记录在您的病历上。研究者、伦理委员会和药品监督管理部门将被允许查阅您的医疗记录。任何有关本项研究结果的公开报告将不会披露您的个人身份。我们将在法律允许的范围内,尽一切努力保护您个人医疗资料的隐私。

可以自愿选择参加研究和中途退出研究

是否参加研究完全取决于您的意愿。您可以拒绝参加此项研究,或在研究过程中的任何时间退出本研究,这都不会影响您和医生间的关系,都不会影响对您的医疗或有其他方面利益的损失。

出于对您的最大利益考虑, 医生或研究者可能会在研究过程中随时中止您继续参加本项研究。

如果您因为任何原因从研究中退出,您可能被询问有关您使用试验药物的情况。如果医生认为需要,您也可能被要求进行实验室检查和体格检查。

#### 9. 受试者声明

受试者签名 , 日期: 年 月 日 联系电话: 受试者家长或监护人签名(只限年龄在 18 岁以下的未成年病人或不能自我表达意见的成年病人): , 日期: 年 月 日 医生姓名(全名): 联系电话: 医生签名: , 日期: 年 月 日 (知情同意书一式两份,医生和受试者各保存一份)